CLINICAL TRIAL: NCT03019835
Title: Can we Antagonize Mivacurium With Neostigmine
Brief Title: Can we Antagonize Mivacurium With Neostigmine ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, JOHN NICOLARDOT, MD, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: B406201629996; U1111-1190-7993 (Other: WHO-UTN)
Record Dates: First submitted 2016-12-22; First posted 2017-01-13 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Mivacurium; Neostigmine; Residual Paralysis
Keywords: mivacurium; neostigmine; antagonism
MeSH Terms: interventions — Neostigmine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- GROUP 1 (Active Comparator): A group receiving neostigmine (40 mcg / kg) when the block Neuromuscular block's recovery measured by acceleromyography is 1 response of 4 in TOF mode (Train Of Four)
  Interventions: Drug: Neostigmine (40 mcg / kg) at different time of neuromuscular block's recovery
- GROUP 2 (Active Comparator): A group receiving neostigmine (40 mcg / kg) when the block Neuromuscular block's recovery measured by acceleromyography is 2 response of 4 in TOF mode (Train Of Four)
  Interventions: Drug: Neostigmine (40 mcg / kg) at different time of neuromuscular block's recovery
- GROUP 3 (Active Comparator): A group receiving neostigmine (40 mcg / kg) when the block Neuromuscular block's recovery measured by acceleromyography is 3 response of 4 in TOF mode (Train Of Four)
  Interventions: Drug: Neostigmine (40 mcg / kg) at different time of neuromuscular block's recovery
- GROUP 4 (Active Comparator): A group receiving neostigmine (40 mcg / kg) when the block Neuromuscular block's recovery measured by acceleromyography is 4 response of 4 in TOF mode (Train Of Four)
  Interventions: Drug: Neostigmine (40 mcg / kg) at different time of neuromuscular block's recovery
- CONTROL (Active Comparator): A control group : not receiving an antagonist (spontaneous recovery)
  Interventions: Other: Spontaneous recovery

INTERVENTIONS:
Drug: Neostigmine (40 mcg / kg) at different time of neuromuscular block's recovery
  Arms: GROUP 1; GROUP 2; GROUP 3; GROUP 4
Other: Spontaneous recovery — just measuring the Train Of Four at 3 6 9 12 and 15 minutes and measure the Train Of Four Ratio
  Arms: CONTROL

SUMMARY:
The antagonism of neuromuscular blocking agents (NMBA) (or curares), as well as the antagonism of other drugs used in anesthesia, is a major challenge for the speciality.

Residual paralysis is indeed a risk factor for post-operative morbidity and mortality and antagonization of curares at the end of the procedure is associated with a reduction in mortality .

Its use should be as large as possible and its contraindications are extremely rare.

The antagonism of the NMBA reduces the duration of the neuromuscular block and the complications that are associated .

In this study, the investigators use mivacurium (or Mivacron) as non-depolarizing curare and neostigmine as an antagonist.

Neostigmine reduces the duration of the neuromuscular block induced by mivacurium, By reducing the breakdown of acetylcholine, neostigmine induces an increase in acetylcholine in the synaptic cleft which competes for the same binding site as nondepolarizing neuromuscular blocking agents, and reverses the neuromuscular blockade.

But the use of neostigmine in current practice is not very widespread in this clinical situation.

The reduction in the duration of the block is significant in comparison with a spontaneous recovery .

Moreover, spontaneous recovery is not always complete and sometimes very long.

Nevertheless, its action is effective and this study could support this use but also specify the duration and the quality of the return to normal of the neuromuscular transmission.

ELIGIBILITY:
Inclusion Criteria:

* Patients American Society of Anesthesiologists (ASA) 1 to 3
* Absence of neuromuscular disease, renal and hepatic insufficiency
* Absence of medication that could interfere with the mediators of the neuromuscular junction

Exclusion Criteria:

* Bronchial asthma
* Parkinson disease
* BMI> 35
* Known hypersensitivity to neostigmine or to any of the excipients of Neostigmine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04-22 (Actual); Study Completion 2017-04-22 (Actual)

PRIMARY OUTCOMES:
Change in TOF ( Train Of Four) measure | for each patient, measure of Train Of Four at 3, 6, 9, 12, 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Michel Baurain, Bruxelles Capitale, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Baurain MJ, Dernovoi BS, d'Hollander AA, Hennart DA. Comparison of neostigmine-induced recovery with spontaneous recovery from mivacurium-induced neuromuscular block. Br J Anaesth. 1994 Dec;73(6):791-4. doi: 10.1093/bja/73.6.791. PMID 7880668
- [Result] Baillard C, Clec'h C, Catineau J, Salhi F, Gehan G, Cupa M, Samama CM. Postoperative residual neuromuscular block: a survey of management. Br J Anaesth. 2005 Nov;95(5):622-6. doi: 10.1093/bja/aei240. Epub 2005 Sep 23. PMID 16183681
- [Result] Szenohradszky J, Fogarty D, Kirkegaard-Nielsen H, Brown R, Sharma ML, Fisher DM. Effect of edrophonium and neostigmine on the pharmacokinetics and neuromuscular effects of mivacurium. Anesthesiology. 2000 Mar;92(3):708-14. doi: 10.1097/00000542-200003000-00015. PMID 10719950
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pubmed/7880668